CLINICAL TRIAL: NCT05689827
Title: Prospective Multicentre Comparative Randomized Double Blind Placebo Controlled Study of Safety and Efficacy of the Therapy With BRAINMAX® for the Treatment of Patients With Asthenia After Having the Novel Coronavirus Infection (COVID-19)
Brief Title: Safety and Efficacy of the Therapy With BRAINMAX® for the Treatment of Patients With Asthenia After COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BRAINMAX_ 2021
Record Dates: First submitted 2023-01-18; First posted 2023-01-19 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Asthenia; COVID-19
MeSH Terms: conditions — Asthenia; COVID-19 | interventions — 3-(2,2,2-trimethylhydrazine)propionate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethyl methyl hydroxypyridine succinate + Meldonium (Experimental): Arm 1 (n=80) received intramuscularly with the dosage regimen of 5 mL of solution (500 mg of ethyl methyl hydroxypyridine succinate + 500 mg of meldonium) once per day for 10 days; total number of injections for the treatment course is 10 and then orally with the dosage regimen of 2 capsules (500 mg of ethyl methyl hydroxypyridine succinate + 500 mg of meldonium) twice per day for 30 days; total number of capsules for the treatment course is 120. Second group received Placebo in the same way.
  Interventions: Drug: Ethyl methyl hydroxypyridine succinate + Meldonium
- Placebo (Placebo Comparator): Arm 2 (n=80) received Placebo in the same way.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ethyl methyl hydroxypyridine succinate + Meldonium — Ethyl methyl hydroxypyridine succinate 100.0 mg/mL, meldonium dihydrate - 100.0 mg/mL (Solution for intravenous and intramuscular administration), then Ethyl methyl hydroxypyridine succinate - 250.0 mg, meldonium dihydrate based on dihydrate without adsorption moisture - 250.0 mg (oral capsules)
  Other Names: BRAINMAX®
  Arms: Ethyl methyl hydroxypyridine succinate + Meldonium
Drug: Placebo — Placebo was used in the same way
  Arms: Placebo

SUMMARY:
This is prospective multicentre comparative randomized double blind placebo controlled study conducted in 6 medical facilities.The objective of the study is to assess the safety and efficacy of the sequential therapy with BRAINMAX®, solution for intravenous infusion and intramuscular injection, and BRAINMAX®, capsules for the treatment of patients with asthenia after having the novel coronavirus infection (COVID-19)

DETAILED DESCRIPTION:
Upon signing the informed consent form and screening, 160 eligible patients from 18 to 65 years of age with asthenia after having the novel coronavirus infection (COVID-19) were randomized at a 1:1 ratio. First group received intramuscularly with the dosage regimen of 5 mL of solution (500 mg of ethyl methyl hydroxypyridine succinate + 500 mg of meldonium) once per day for 10 days; total number of injections for the treatment course is 10 and then orally with the dosage regimen of 2 capsules (500 mg of ethyl methyl hydroxypyridine succinate + 500 mg of meldonium) twice per day for 30 days; total number of capsules for the treatment course is 120. Second group received Placebo in the same way.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to sign the patient informed consent form for the participation in the clinical study
2. Patients of both sexes of 18-65 years of age
3. Patient's negative test result for severe acute respiratory syndrome (SARS) -CoV-2 RNA obtained by polymerase chain reaction (PCR) method within 72 hours
4. COVID-19 diagnosis documented in the history more than 12 weeks ago*
5. Minimum two symptoms of asthenic state: fatigue, atony, dizziness, sleeping disorder, feeling of energy loss and decreased functioning, intellectual function disorder, attention and memory disorder, which appeared during or after COVID-19, retain for more than 12 weeks and cannot be explained by an alternative diagnosis
6. Patients capable of following the requirements of the Clinical Study Protocol
7. Negative pregnancy test result (for women with the active childbearing potential)
8. MFI-20 scale score is more than 30 at the moment of screening.

Exclusion Criteria:

1. Allergic reactions to the components of the study product
2. Oxygen saturation by pulse oximetry (SpO2) oxygen saturation ≤ 95%
3. Depression level score by Hamilton Depression Rating Scale (HDRS) at the screening ≥ 8
4. Intracranial pressure rise (for the reason of venous outflow disorder and intracranial tumours)
5. Severe hepatic failure
6. Severe renal failure
7. Chronic liver and hepatic diseases
8. Thyroid diseases
9. Anaemia
10. Malignant tumour of any localization currently or during 5 years before the inclusion into the study except for completely treated carcinoma in situ
11. Autoimmune diseases
12. Other chronical diseases which, according to the investigator, can cause asthenia
13. G lomerular filtration rate (GFR) parameter at screening < 30 mL/min
14. Pregnancy or lactation period
15. Participation in any other clinical study during the last 3 months
16. Tuberculosis, cancers or positive reaction to the HIV infection, hepatitis B & C, syphilis according to the history data
17. Severe eyesight and/or hearing disorders, serious articulation disorders and/or other deviations able to prevent the patient from adequate cooperation during the study)
18. Mental disorders in the history
19. Alcohol, drug abuse or drug dependence in the history
20. Patients which, according to the investigator, are obviously or probably incapable of understanding and evaluating this study information within the process of the informed consent form signing, including but not limited to with regard to expected risks and possible discomfort
21. Other diseases, symptoms or conditions not listed above, which, according to the investigator, are predicaments for the participation in the clinical study

Exclusion of patients from the study

1. Erroneous inclusion (inclusion and exclusion criteria violation).
2. Investigator or Sponsor's decision to exclude the patient from the study because of clinically significant deviation from protocol/protocol violation.
3. Serious adverse events or adverse events which do not meet the seriousness criteria and which if developed, according to the investigator, can make the patient's further participation in the study harmful for the patient's health or wellbeing.
4. Any adverse event (there might be no connection with the study drug intake) requiring the observation, procedures and/or drug treatment not allowed by this study protocol.
5. Patient's refusal to continue the participation in the study or his/her lack of discipline.
6. Allergic reaction to the study drug intake, which require its discontinuation.
7. Patient's wish to prematurely terminate the study for any reason.
8. Loss of contact with the patient and his/her absence for the visit.
9. Necessity to use a therapy prohibited by this protocol.
10. Occurrence of pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Asthenia on a scale Multidimensional Fatigue Inventory (MFI-20) after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Mean decrease of MFI-20 asthenia scale score after the completion of the sequential therapy

SECONDARY OUTCOMES:
Asthenia on a scale MFI-20 after the completion of the parenteral therapy | From baseline to Visit 3 (day 11)
  Mean decrease of MFI-20 asthenia scale score after the completion of the parenteral therapy
Asthenia on a scale MFI-20 after the completion of the oral therapy | From Visit 3 (day 11) to Visit 5 (day 41)
  Mean decrease of MFI-20 asthenia scale score after the completion of the oral therapy
Headache on a visual analogue scale (VAS) after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Score dynamics by VAS for the headache evaluation after the completion of the sequential therapy
Headache on a VAS after the completion of the parenteral therapy | From baseline to Visit 3 (day 11)
  Score dynamics by VAS for the headache evaluation after the completion of the parenteral therapy
Headache on a VAS after the completion of the oral therapy | From Visit 3 (day 11) to Visit 5 (day 41)
  Score dynamics by VAS for the headache evaluation after the completion of the oral therapy
Sleep Quality on a Pittsburgh sleep quality index (PSQI) after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Score dynamics by PSQI questionnaire after the completion of the sequential therapy
Fatigue on a Fatigue Assessment Scale (FAS-10) scale after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Score dynamics by FAS-10 scale after the completion of the sequential therapy
Fatigue on a FAS-10 scale after the completion of the parenteral therapy | From baseline to Visit 3 (day 11)
  Score dynamics by FAS-10 scale after the completion of the parenteral therapy
Fatigue on a FAS-10 scale after the completion of the oral therapy | From Visit 3 (day 11) to Visit 5 (day 41)
  Score dynamics by FAS-10 scale after the completion of the oral therapy
Dizziness on a Dizziness Handicap Inventory (DHI) questionnaire after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Score dynamics by DHI questionnaire after the completion of the sequential therapy
Dizziness on a DHI questionnaire after the completion of the parenteral therapy | From baseline to Visit 3 (day 11)
  Score dynamics by DHI questionnaire after the completion of the parenteral therapy
Dizziness on a DHI questionnaire after the completion of the oral therapy | From Visit 3 (day 11) to Visit 5 (day 41)
  Score dynamics by DHI questionnaire after the completion of the oral therapy
Cognitive function on a Monreal Gognitive Assessment (MoCA) scale after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Score dynamics by MoCA scale after the completion of the sequential therapy
Anxiety on a Beck scale after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Score dynamics by Beck scale after the completion of the sequential therapy
Anxiety on a Beck scale after the completion of the parenteral therapy | From baseline to Visit 3 (day 11)
  Score dynamics by Beck scale after the completion of the parenteral therapy
Anxiety on a Beck scale after the completion of the oral therapy | From Visit 3 (day 11) to Visit 5 (day 41)
  Score dynamics by Beck scale after the completion of the oral therapy
Regulatory function on a Kerdo vegetation index after the completion of the sequential therapy | From baseline to Visit 5 (day 41)
  Changes in values of Kerdo vegetation index after the completion of the sequential therapy
Regulatory function on a Kerdo vegetation index after the completion of the parenteral therapy | From baseline to Visit 3 (day 11)
  Changes in values of Kerdo vegetation index after the completion of the parenteral therapy

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Federal State Budgetary Research Institution "Research Centre of Neurology", Moscow
  - OsteoVita LLC, Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "Municipal Hospital No. 40 of Kurortny District", Sestroretsk
  - Centre For Evidence-Based Medicine Llc, Yaroslavl
  - Medical Centre of Diagnostics and Prevention Plus LLC, Yaroslavl
  - State Budgetary Healthcare Institution of Yaroslavl Region "Yaroslavl Region Clinical Hospital for War Veterans - International Elderly People Centre 'Zdorovoe Dolgoletie', Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanashyan MM, Raskurazhev AA, Kuznetsova PI, Bely PA, Zaslavskaya KI. [Prospects and possibilities for the treatment of patients with long COVID-19 syndrome]. Ter Arkh. 2022 Dec 26;94(11):1285-1293. doi: 10.26442/00403660.2022.11.201981. Russian. PMID 37167167
- See also: Cyberleninka is an open access scientific electronic library — https://cyberleninka.ru/article/n/perspektivy-i-vozmozhnosti-terapii-patsientov-s-astenicheskim-sindromom-posle-perenesennoy-novoy-koronavirusnoy-infektsii-covid-19